CLINICAL TRIAL: NCT03510988
Title: Dedicated Breast PET/MRI in Evaluation of Extent of Disease in Women With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily paused per study team for interim data review.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1705018188
Record Dates: First submitted 2018-04-05; First posted 2018-04-27 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Newly Diagnosed Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Women with newly diagnosed breast cancer (Experimental): Women with newly diagnosed breast cancer recruited for hybrid dedicated breast PET/MRI for extent of disease staging prior to management in lieu of breast MRI alone. IV FDG and Gadolinium was injected once prior to the study as per protocol and weight. In each second consecutively recruited patient FDG dosage was decreased by 20% up to 40% of weight-based dosage to ascertain feasibility of imaging at lower FDG dosages. IV Gadolinium was injected once with weight dependent dosages as per clinical standard of care.
  Interventions: Diagnostic Test: Hybrid breast FDG PET/MRI

INTERVENTIONS:
Diagnostic Test: Hybrid breast FDG PET/MRI — Hybrid breast FDG PET/MRI

SUMMARY:
This is a single institution study enrolling women over age 25 with newly diagnosed breast cancer and for whom a breast MR has been ordered as standard of care. Subjects will undergo a hybrid dedicated Breast PET/MRI in lieu of a breast MRI alone, for evaluation of extent of disease prior to surgical and oncologic management. The study will investigate any incremental added benefit to breast MRI specificity by the addition of concurrent hybrid breast PET.

DETAILED DESCRIPTION:
The study hypothesis is that the combination of Breast PET/MRI, will improve specificity and decrease the number of false positive breast biopsies recommended based on breast MRI findings.

ELIGIBILITY:
Inclusion Criteria:

* Women over age of 25 with newly diagnosed breast cancer and for whom a breast MR has been ordered as standard of care

Exclusion Criteria:

* Male subjects
* Women younger than 25
* Pregnant subjects
* Unable or unwilling to undergo MRI
* Previous adverse reaction to 18F-FDG
* Unwilling to undergo biopsy of MRI positive lesions

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Dodelzon, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With Newly Diagnosed Breast Cancer
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Specificity of the PET-MRI Compared to MRI Alone as Assessed by the Percentage of True Negatives Out of All Benign/Non-malignant Lesions Breast Cancer
Description: Blinded breast imaging readers were provided at random a reading list of anonymized studies of breast PET/MRIs and MRI alone from the study cohort and asked to assess lesions suspicious for malignancy. Specificity of all lesions on PET-MRI compared to MRI alone is assessed by the percentage of true negatives out of all benign/non-malignant lesions.
Time Frame: 24 months
Measure: Number (90% Confidence Interval); unit: percentage of true negative
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 14
percentage of true negative
  Specificity of MRI alone | 63.89 [59.1 to 68.9]
  Specificity of PET-MRI | 83.33 [74.9 to 91.1]

2. Secondary Outcome: Sensitivity, PPV (Positive Predictive Value), and NPV (Negative Predictive Value) for the Diagnosis Based on the Entire PET/MRI and MRI Alone Will be Calculated and Reported Along With the Corresponding Two-sided 90% Confidence Intervals.
Description: Blinded radiologists evaluated a list of anonymized studies of breast MRI alone and after washout period the same MRI with ovelayed PET from a hybrid PETMRI study cohort and asked to assess lesions suspicious for malignancy in addition to known index tumor. Measures of diagnostic accuracy( sensitivity, specificity, PPV and NPV) for any and all additional lesions exclusive of the known index tumor detected by readers were calculated for MRI alone and for PET/MRI. Due to washout period readers assessed the imaging of hybrid PET/MRI in complement, as such readers may assess previously questioned MRI findings as benign in the absence of FDG uptake. Sensitivity is the % of true positive & specificity is the % of true negative. PPV is the probability that if imaging was assessed as suspicious on biopsy was malignant. NPV is the % likelihood that if imaging was assessed as negative there was no additional malignancy on surgical excision.
Time Frame: 24 months post-intervention
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 14
percentage
  Sensitivity of MRI alone | 66.67 [39.6 to 94.4]
  Sensitivity of PET-MRI (percent true positives exclusives of the index tumor) | 0 [0 to 0]
  PPV of MRI alone | 23.53 [18.1 to 27.9]
  PPV of PET-MRI(% probability of true positives exclusive of the index tumor) | 0 [0 to 0]
  NPV of MRI alone | 92.00 [86.6 to 98.7]
  NPV of PET-MRI | 83.33 [81.5 to 84.5]

3. Secondary Outcome: Average Signal to Noise Ratios (SNR) vs. IV FDG Dosages Will be Summarized in Plot Format.
Description: PET imaging was assessed for signal-to-noise ratio of maximum standardized uptake value (SUVmax) over the breast background SUVmean. This is compiled below for each administered dose of FDG. Each subject received one FDG and one gadolinium dose IV injection.
Time Frame: 24 months post-intervention
Population: The average signal to noise ratio was unable to be measured for one subject.
Measure: Mean (Standard Deviation); unit: average signal to noise ratio
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 13
average signal to noise ratio
  Dose Proportion of standard 10 mCi IV FDG dose: 1.01: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 1.01 | 1.799
  Dose Proportion of standard 10 mCi IV FDG dose: 1.007: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 1.007 | 4.427
  Dose Proportion of standard 10 mCi IV FDG dose: 0.802: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.802 | 9.333
  Dose Proportion of standard 10 mCi IV FDG dose: 0.805: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.805 | 2
  Dose Proportion of standard 10 mCi IV FDG dose: 0.6: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.6 | 6.25
  Dose Proportion of standard 10 mCi IV FDG dose: 0.631: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.631 | 4
  Dose Proportion of standard 10 mCi IV FDG dose: 0.505: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.505 | 5.222
  Dose Proportion of standard 10 mCi IV FDG dose: 0.491: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.491 | 13.3
  Dose Proportion of standard 10 mCi IV FDG dose: 0.58: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.58 | 11.333
  Dose Proportion of standard 10 mCi IV FDG dose: 0.65: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.65 | 6.778
  Dose Proportion of standard 10 mCi IV FDG dose: 0.593: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.593 | 4.6
  Dose Proportion of standard 10 mCi IV FDG dose: 0.4: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.4 | 3.2
  Dose Proportion of standard 10 mCi IV FDG dose: 0.401: number analyzed (Participants) | 1
  Dose Proportion of standard 10 mCi IV FDG dose: 0.401 | 11

4. Secondary Outcome: Number of Interval Recurrences
Time Frame: 24 months post-intervention
Measure: Number; unit: participants
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 14
participants | 1

5. Secondary Outcome: Sensitivity in Detection of Axillary and Internal Mammary Lymph Node Metastasis Between the Hybrid Breast FDG PET/MRI vs Breast MRI Alone Will be Summarized
Description: Blinded breast imaging readers were provided at random a reading list of anonymized studies of breast PET/MRIs and MRI alone from the study cohort and asked to assess nodal disease as a whole (present/absent). Sensitivity, specificity, PPV (positive predictive value), and NPV (negative predictive value) of nodal metastasis (presence or absence) of hybrid breast FDG PET/MRI vs breast MRI alone were compared. Due to washout period readers assessed the imaging of hybrid PET/MRI in complement, as such readers may assess previously questioned MRI findings as benign in the absence of FDG uptake.
Time Frame: 24 months post-intervention
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 14
percentage
  Sensitivity of MRI alone | 33.33 [-21.8 to 87.8]
  Sensitivity of PET-MRI ( percent of true positive nodal disease in addition to MRI alone) | 0 [0 to 0]
  Specificity of MRI alone | 76.92 [57.8 to 96.2]
  Specificity of PET-MRI | 87.18 [78.8 to 95.2]
  PPV of MRI alone | 10.00 [-21.8 to 87.8]
  PPV of PET-MRI (% probability of true positives of nodal disease) | 0 [0 to 0]
  NPV of MRI alone | 93.75 [87.2 to 98.8]
  NPV of PET-MRI | 91.89 [91.5 to 92.5]

6. Secondary Outcome: Perceived Patient Benefit of Undergoing a Simultaneous FDG PET/MRI Will be Summarized
Description: Subjects will be asked to fill out a questionnaire at the conclusion of their breast PET/MRI exam assessing on a scale of 1 - 5 how important it was for them to save time to do the PET/MRI simultaneously knowing that they may have a negative PET/MRI for extent of disease (no additional sites of disease aside from index cancer), how valuable it is for them to potentially avoid unnecessary biopsies if the study hypothesis is correct, and how important it is to them to decrease delay to surgery.
Time Frame: 24 months post-intervention
Population: Seven out fourteen subjects elected to complete the questionnaire.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Women With Newly Diagnosed Breast Cancer
Number analyzed (Participants) | 7
scores on a scale | 4.28 (0.49)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Women With Newly Diagnosed Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Wilson method was not utilized for the confidence intervals for multiple outcome measures at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT03510988/Prot_SAP_000.pdf